CLINICAL TRIAL: NCT03703986
Title: Explore the Causes and Predictors of Early Neurological Deterioration Occurred in Patients With Acute Ischemic Stroke
Brief Title: Early Neurological Deterioration in Patients With Acute Ischemic Stroke
Acronym: ENDAIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-SR-099
Record Dates: First submitted 2018-06-26; First posted 2018-10-12 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Infarction
Keywords: deterioration; risk factors; predictors
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- END group: The patients in this group had an elevation of ≥ 2 points in the National Institute of Health Stroke Scale (NIHSS) within 7 days of stroke onset.
- non-END group: The patients in this group had a slight increase of < 2 points or a decrease in NIHSS within 7 days of stroke onset.

SUMMARY:
This study set out to explore the risk factors of early neurological deterioration (END) occurred in patients with acute ischemic stroke and to investigate the corresponding predictors.

DETAILED DESCRIPTION:
END refers to the illness aggravation occurred in the early stage of stroke and often indicates a poor outcome. Some clinical scales may play an important role in its diagnoses and treatments. Across the reviewed studies, the risk factors of END, which included biochemical parameters, neuroimaging, ect. were explored incompletely and the effective predictors of END is unknown. We aimed to explore the risk factors of END and investigate the predictive value of certain scales.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute ischemic stroke
* Subjects with detailed progress notes

Exclusion Criteria:

* Subjects with thrombolysis therapy
* Subjects with transient ischemia attach
* Subjects complicated with seriously underlying diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to First Affiliated Hospital of Nangjing Medical University from January 2015 to April 2018 were collected retrospectively.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale | 7 days
  National Institutes of Health Stroke Scale (NIHSS) can assess the severity of stroke. The total score of NIHSS ranges from 0 to 42, with higher scores indicating better neurological function.
Canadian Neurological Scale | 7 days
  Canadian Neurological Scale (CNS) can assess the severity of stroke as well. The total score of CNS ranges from 0 to 10, with higher scores indicating worse neurological function.

SECONDARY OUTCOMES:
Blood parameters | 7days
  The blood parameters included total cholesterol, triglyceride, low-density lipoprotein and high-density lipoprotein. The normal range of them were 3 mmol·L-1 to 5.7 mmol·L-1, 0 mmol·L-1 to 2.25 mmol·L-1, 2.6 mmol·L-1 to 4.1 mmol·L-1, 1.03 mmol·L-1 to 1.55 mmol·L-1, respectively.
Neuroimaging data | 7days
  Intracranial stenosis was defined as ≥ 50% narrowing in any of the intracranial arteries. Multi-vessel lesions were recorded when the number of cerebral vascular stenosis was greater than 2.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, China